CLINICAL TRIAL: NCT07316582
Title: Clinical and Biochemical Evaluation of Melatonin Loaded in Injectable Platelet-Rich Fibrin in the Management of Stage II Grade A Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Melatonin Loaded in Injectable Platelet-Rich Fibrin in the Management Periodontitis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Nora Abdelgawad Mohamed, Associate Professor of Oral Medicine, Periodontology and Diagnosis, Faculty of Dental Medicine for girls, Al -Azhar University, Cairo, Egypt, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-ME-25-16
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis Stage II
MeSH Terms: conditions — Periodontitis | interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scaling and Root Planning only (No Intervention): Mechanical removal of supra- and subgingival plaque and calculus using ultrasonic and hand instruments.
- Injectable Platelet-Rich Fibrin (i-PRF) (Placebo Comparator): local application of injectable platelet-rich fibrin (i-PRF) into periodontal pockets.
  Interventions: Biological: injectible platelet rich fibrin (i-PRF )
- scaling and Root Planing plus Melatonin-Loaded Injectable Platelet-Rich Fibrin (Experimental): patients will be included in this group receiving SRP with Melatonin loaded in (I-PRF) using insulin syringe for injection
  Interventions: Drug: Melatonin-Loaded Injectable Platelet-Rich Fibrin

INTERVENTIONS:
Drug: Melatonin-Loaded Injectable Platelet-Rich Fibrin — patients will be included in this group receiving SRP with Melatonin loaded in (I-PRF) using insulin syringe for injection
  Arms: scaling and Root Planing plus Melatonin-Loaded Injectable Platelet-Rich Fibrin
Biological: injectible platelet rich fibrin (i-PRF ) — patients will be included in this group receiving (SRP) with local application of i-PRF
  Arms: Injectable Platelet-Rich Fibrin (i-PRF)

SUMMARY:
melatonin loaded in injectible platelet rich fibrin in treatment of periodontitis

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with stage II periodontitis based on AAP/EFP 2018 classification

• Minimum of two non-adjacent periodontal pockets <5 mm in different quadrants

• Systemically healthy individuals willing to participate and comply with follow-up visits

• Radiographic bone loss (ranged from is 10-20% mostly horizontal

Exclusion Criteria:

History of systemic diseases affecting periodontium (e.g., diabetes, osteoporosis)

• Use of antibiotics, anti-inflammatories, or antioxidant supplements in the past 3 months

• Smoking or tobacco use

• Pregnancy or lactation

• Allergy to melatonin or related compounds

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine for girls Al-Azhar University, New Cairo, Egypt